CLINICAL TRIAL: NCT02895724
Title: Hyperbaric Oxygen Therapy to Reduce Lymphedema After Breast Cancer -an Explorative Clinical Trial
Acronym: HBOT-LYCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Oksbjerg Dalton, MD PhD, Danish Cancer Society
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-16019587
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Secondary Lymphedema
Keywords: Hyperbaric oxygen therapy; secondary lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBOT receivers (Experimental): Participants in a post breast cancer surgery randomized controlled trial detected with lymphedema 1 year postoperatively are invited to 40 consequtive treatments of hyperbaric oxygen therapy to reduce lymphedema. The experimental drug is 100% medical oxygen given in a pressure chamber of 2,4 bar,every treatment lasting approximately 100 minutes.
  Interventions: Drug: Medical Oxygen
- blodsample comparison (No Intervention): Matched Lymphedema free participants from LYCA Exercise recruited to donate blood samples for comparison on important blod biomarkers and collagen levels.

INTERVENTIONS:
Drug: Medical Oxygen — Hyperbaric oxygen therapy
  Arms: HBOT receivers

SUMMARY:
The purpose of this study is to examine if pressurechamber treatment (HBOT) can reduce early stages of breast cancer related lymphedema, and to explore the mechanisms involved in the disease progress.

DETAILED DESCRIPTION:
Lymphedema (LE) is a potential complication of primary breast cancer treatment and the influence of LE on the quality of life is well-established. To date there is no established treatment that can reverse lymphedema. Patients are dependent on compression garments and manual lymphatic drainage to prevent progression of LE and worsening of discomfort, pain, upper limb dysfunction/sensation, skin problems and infections.

As a development in treatment of tissue damage after radiation treatment HBOT is used in the treatment of radiation induced mandibular necrosis, hemorrhagic cystitis or proctitis following pelvic radiation. The pathology, which correlates to the effect of HBOT include neovascularization, as well as organization and reduction in fibrous tissue, and new evidence also shows an increase in the number of lymphatic vessels in irradiated oral mucosa. Some studies have found that HBOT might also reduce arm edema in breast cancer patients, but evidence is inconsistent and mainly based on chronic and long existing lymphedema in long term BC survivors. The investigators argue that the possibility of remodeling of mature fibrotic tissue is less pronounced when the lymphedema has been present over prolonged periods of years, limiting the possibility of treatment success. Although HBOT is a lengthy and time-consuming treatment, it is documented safe in all aspects with little risk of side effects, and the potential health gains from the treatment are immense.

This explorative HBOT trial was designed to generate hypotheses about the conditions under which HBOT is effective to reduce lymphedema, and to reveal new aspects of the role of tissue composition on the effectiveness of HBOT. The early initiation of HBOT is the key factor in this set up, which is different from the previous studies in the field. To be able to do so, all participants in a randomized controlled exercise trial (LYCA), who develop lymphedema during the first year after surgery will be invited to participate in the HBOT trial.

This trial was accepted with regards to the experimental use of medical oxygen in a pressure chamber for the treatment of lymphedema in the National Health and Medicines Authority in 2015; protocol number R96- A6604-14- S22, EUDRACT no: 2015-000604-25.

Aims and hypothesis The primary aim in this explorative trial is to examine whether HBOT is effective in treating early LE. Secondly, the aim is to examine the importance of the conditions under which HBOT is more effective in treating LE. Effects of HBOT (primary endpoints) will be evaluated as objective measurements of the affected and contralateral arm volume assessed by DXA scan and Light perometry. Changes in lymphatic clearance rate before and after HBOT (secondary endpoint) will be measured by lymphoscintigraphy and biomarkers of inflammation and collagen levels in blood samples. Other secondary endpoints are patient reported outcomes of symptoms of lymphedema, physical and psychological function, fatigue, and quality of life, and will be assessed by questionnaire.

It is hypothesized that HBOT will reduce the volume and symptoms of persistent LE in the patients receiving this treatment, to a clinically non-significant level. Furthermore, it is hypothesized that HBOT cause reduced patient reported symptoms of lymphedema and fatigue and increased physical and psychological function and quality of life.

Method

The LYCA HBOT trial is an explorative and observational study, offering all participants in the exercise trial, who develop lymphedema, a treatment course with HBOT. In addition, an equal number of matched control subjects without lymphedema from the exercise trial will be included for blood sampling and DXA scans. It is planned to start in September 2016 and to be ended with the last follow up (6 months) of the last participant, in May 2018. Patients are invited at 12 months follow-up in the LYCA exercise trial if they present with the following criteria for lymphedema persisting more than 4 weeks:

* a swelling of the arm on the operated side, corresponding to >3% increase in inter limb volume change from the baseline measurement
* a score of 2 points or more on numeric rating scale for self reported swelling, heaviness and tightness
* a clinical exam where 2 or more of the following 4 criteria must be present (i-iii are compared with the unaffected side): i) decreased visibility of subcutaneous veins on the ventral lower arm or dorsal hand ii) loss of normal contours in the region of the medial side of the elbow/distal end of the upper arm iii) thicker skin and subcutis on palpation iv) pitting edema

The HBOT component:

HBOT includes compression to 2.4 Bar (ATA) in a multi-place hyperbaric chamber at Rigshospitalet. Patients breathe 100% oxygen via a transparent hood for a total of 100 minutes including two 5-minutes periods of de- and ascent. The course of treatment comprises a total of 40 pressure exposures, distributed as 5 days a week for 8 continuous weeks. The women will be encouraged to continue exercising 3 times a week throughout the treatment period, adherence to exercise promoted by mobile phone text messages.

Analysis For this explorative trial, no power calculation is carried out, due to the explorative focus to generate hypotheses. Descriptive statistics will be used to look at possible tendencies, associations and differences. Arm volume over time will be compared, and limb volume difference in those women who have carried out the progressive resistance training compared to the women who received the usual care control condition will be evaluated. Furthermore, the possible association between effect of HBOT and amount of exercise will be examined, as will the increase in or level of muscle strength, symptom burden, body composition, physical function, and health related quality of life.

In analysis of blood samples of HBOT participants and control subjects, levels of the biomarkers in question will be compared and contrasted, both at baseline (before HBOT) and in changes over time (during and after HBOT). Within the groups of controls and HBOT participants, there are individuals from each LYCA-exercise intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Participant in "LYCA - exercise"
* Declared cancer free
* Completed chemotherapy and radiotherapy (maximum 1 year after completed treatment)
* Lymphedema present when measured at "Lyca-exercise" 1 year follow-up: >3% increase in inter limb volume change from the baseline measurement, AND a score of 2 points or more on NRS for symptoms (heaviness, tightness, swelling), persisting more than 4 weeks
* Two or more of the following clinical criteria must be present (i-iii are compared with the unaffected side): i) decreased visibility of subcutaneous veins on the ventral lower arm or dorsal hand, ii) loss of normal contours in the region of the medial side of the elbow/distal end of the upper arm, iii) thicker skin and subcutis on palpation, iv) pitting edema.

Exclusion Criteria

* Pregnancy
* Undrained pneumothorax
* Unability to equalize pressure in the ears in spite of drain treatment by Ear- Nose- and Throat specialist.
* Severe heart failure detected during pre-examination for HBOT
* Intractable Claustrophobia non-responsive of standard pre-medication

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Arm volume | 8 months
  measured by perometry and DXA scans

SECONDARY OUTCOMES:
lymph clearance | 8 months
  upper limb lymph clearance rate measured by quantitative lymphoscintigraphy
Functional impairment | 8 months
  upper limb functional impairment measured by queationnaire: "Lymph ICF"
psychological well-being | 8 months
  anxiety, depression and health realted quality of life measured by questionnaire
blood biomarkers | 8 months
  biomarkers of inflammation and levels of collagen measured by blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hyldegaard, DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: Undecided